CLINICAL TRIAL: NCT05573009
Title: The Effect of Stress Reduction Program Based on Cognitive Behavioral Approach on Pregnancy Process and Mental Health in High Risk Pregnant Women
Brief Title: The Effect of Stress Reduction Program on Pregnancy Process and Mental Health in High Risk Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nesibe Kalyoncu, PhD Candidate Nurse, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IstanbulU-NKALYONCU-001
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Pregnancy, High Risk; Depression, Postpartum; Anxiety in Pregnancy; Stress Disorder
Keywords: pregnancy, high risk; depression, postpartum; anxiety in pregnancy
MeSH Terms: conditions — Depression, Postpartum; Stress Disorders, Traumatic

STUDY DESIGN:
Intervention Model Description: The study was planned as an experimental study with a randomized control group including pre-test, post-test and follow-up measurements to examine the effect of "stress reduction program based on cognitive behavioral approach" on the maternal mental health, pregnancy, and childbirth process of the high risk pregnant women.
Who Masked: Participant, Care Provider
Masking Description: The women included in the sample of the study do not know which group they are involved in. The data of the experimental and control group was also hidden from the staff of the clinic. One by one interviews were performed in order to prevent the women from contacting each other in the experimental, and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): Five days lasting stress reduction program based on cognitive behavioral approach(each session will be an average of 60 minutes) will be initiated in the third day of hospitalisation to the intervention group.
  At least 3-days of the cognitive behavioral approach-based stress reduction program will be given as face to face interviews to the intervention group during hospitalisation, and the remaining sessions will be given at the bedside as long as the hospitalization continues. If the patient is discharged, the remaining 2 sessions will be completed online.
  Interventions: Behavioral: cognitive behavioral approach-based stress reduction program
- Control Group (No Intervention): Routine nursing care will be provided to the control group along with a stress management manual.

INTERVENTIONS:
Behavioral: cognitive behavioral approach-based stress reduction program — Five days lasting stress reduction program based on cognitive behavioral approach(each session will be an average of 60 minutes) will be initiated in the third day of hospitalisation to the intervention group.
  Session main topics are:
  Session 1 - Introducing the purpose and content of the program - Stress Psychoeducation Session 2 - Cognitive restructuring Session 3 -Behavioral coping Session 4 - Problem solving training Session 5-Upcoming parenthood
  Arms: Training Group

SUMMARY:
Introduction Pregnancy and giving birth to an infant is a physiological process as well as it is also a transition of life, and a stressful period of time with a significance in the life of woman. This period is evaluated as a developmental crisis for the woman, and for her family.

High-risk pregnant women are at the forefront of the individuals who need to be supported the most during the transition to motherhood.The presence of a physiological, emotional and psychosocial condition that endanger the health and life of the pregnant and/or fetus and increases the risk of illness and death is defined as "high-risk pregnancy". Exposure to obstetric complications is known to be associated with the later development of psychiatric disorders.

In the literature review, it is seen that there are few studies in which CBT and mindfulness-based interventions are applied to reduce stress, anxiety and depression in risky or risk-free pregnant women. However, no CBT-based stress reduction program applied to high-risk pregnant women has been found in our country. A stress reduction program based on cognitive behavioral interventions during the transition to motherhood can contribute to the protection of maternal mental health and psychological well-being in pregnant women, and may help for healthy pregnancy and birth outcomes.

Research Aim This study was planned to examine the effect of cognitive behavioral approach-based stress reduction program on pregnancy process and maternal mental health to be applied to high-risk pregnant women.

Research Type The study was planned as an experimental study with a randomized control group including pre-test, post-test and follow-up measurements to examine the effect of "stress reduction program based on cognitive behavioral approach" on the maternal mental health, pregnancy, and childbirth process of the high risk pregnant women.

DETAILED DESCRIPTION:
Introduction Pregnancy and giving birth to an infant is a physiological process as well as it is also a transition of life, and a stressful period of time with a significance in the life of woman. This period is evaluated as a developmental crisis for the woman, and for her family.

High-risk pregnant women are at the forefront of the individuals who need to be supported the most during the transition to motherhood.The presence of a physiological, emotional and psychosocial condition that endanger the health and life of the pregnant and/or fetus and increases the risk of illness and death is defined as "high-risk pregnancy" Exposure to obstetric complications is known to be associated with the later development of psychiatric disorders.

A woman diagnosed with a high-risk pregnancy is experiencing the excitement of becoming a mother despite all the uncertainty, while on the other hand she is trying to cope with important complications such as premature birth risk and infection. During this period, the pregnant woman needs biopsychosocial support. However, in the care management of a high-risk pregnant in hospitals, only the physiological elements can be focused and social, psychological and spiritual care can be ignored.The pregnant woman who cannot meet these requirements, in the postpartum period, it is possible to experience inability to adapt to the maternal role, posttraumatic stress syndrome, postpartum blues or postpartum depression (PPD).

The researchers stated that if the prenatal stress level decreases in depressed women with high-risk pregnancies, the depression indicators will also tend to decrease, and they stated that new psychosocial approaches are needed. Psychotherapeutic interventions are highly effective methods for peripartum depression, anxiety and stress; includes cognitive behavioral therapy (CBT), mindfulness therapy, problem-solving therapy, stress reduction therapy, psychoeducational intervention, or a combination of these.

In the literature review, it is seen that there are few studies in which CBT and mindfulness-based interventions are applied to reduce stress, anxiety and depression in risky or risk-free pregnant women.However, no CBT-based stress reduction program applied to high-risk pregnant women has been found in our country. A stress reduction program based on cognitive behavioral interventions during the transition to motherhood can contribute to the protection of maternal mental health and psychological well-being in pregnant women, and may help for healthy pregnancy and birth outcomes.

Research Aim This study was planned to examine the effect of cognitive behavioral approach-based stress reduction program on pregnancy process and maternal mental health to be applied to high-risk pregnant women.

Research Type The study was planned as an experimental study with a randomized control group including pre-test, post-test and follow-up measurements to examine the effect of "stress reduction program based on cognitive behavioral approach" on the maternal mental health, pregnancy, and childbirth process of the high risk pregnant women.

The target population and sample of the research:

The target population of the research consists of pregnant women hospitalized in the high-risk pregnancy service of a university hospital. The sample of the study was calculated by power analysis using the GPower 3.1.9.7 program. The detected number of the sample was found as 46 including minimum 23 for each group for power: 0.95 when the effect size was taken as 1.25 for identifying the differentiation of score change by the time as a result of the power analysis performed based on a similar study for the research to be designed as one intervention and one control group. Considering the losses that may be experienced during the practice, as many as 50% of the sample group will be included in the study. The experimental group is predicted to include 40 people, and the control group is predicted to include 40 people.

Research Protocol The research will be conducted between March 2022, and March 2023, and will last in a total of 12 months. The research will be conducted in a single center in Istanbul University Istanbul Faculty of Medicine High-Risk Pregnancies (Perinatology) service of the Department of Obstetrics and Gynecology. The detailed study plan is given below.

The study plan:

1. Details of the cognitive behavioral based(CBB) stress reduction program will be created, and expert opinions will be taken.
2. The pilot study and revision of the developed program will be carried out.
3. Pregnant women who meet the research criteria and agree to participate in the study will be assigned to the experimental, and control groups using the randomization method. Randomization of the groups will be performed on a simple random basis using the site www.random.org. Women with high-risk pregnancies will be placed in the experimental and control groups by applying randomization using a simple random number table according to the order of hospitalization in Istanbul University Istanbul Faculty of Medicine.
4. Preliminary interviews will be conducted with the experimental and control groups and the first measurements and data (Information Form, Uncertainty Intolerance Scale, Depression, Anxiety and Stress Scale and Psychological Well-Being Scale) will be collected.
5. Five days lasting stress reduction program based on cognitive behavioral approach(each session will be an average of 60 minutes) will be initiated in the third day of hospitalisation to the intervention group whereas routine nursing care will be provided to the control group along with a stress management manual.
6. At least 3-days of the cognitive behavioral approach-based stress reduction program will be given as face to face interviews to the intervention group during hospitalisation, and the remaining sessions will be given at the bedside as long as the hospitalization continues. If the patient is discharged, the remaining 2 sessions will be completed online.
7. After the intervention program is completed (7th day of hospitalisation), scales will be applied to the intervention and control groups for post-intervention measurements (Uncertainty Intolerance Scale, Depression, Anxiety and Stress Scale and Psychological Well-Being Scale). In addition to the scales, Program Evaluation and Satisfaction Questionnaire will be performed only for the intervention group.
8. After the completion of the program, supportive interviews will be conducted weekly until the childbirth as well as the hospitalisation continues so that the patient can practice the learned data, and once in two weeks on the phone if the patient is discharged from hospital.
9. The week of birth, mode of birth, birth weight, and APGAR scores of the experimental and control group will be recorded from the hospital records.
10. Follow-up measurements will be applied to the intervention and control groups at 4-6 weeks of the postpartum period, and at the end of the third month (Uncertainty Intolerance Scale, Depression, Anxiety and Stress Scale and Psychological Well-Being Scale, Edinburgh Postpartum Depression Scale). After the program is completed, cognitive-behavioral approach based stress reduction program will be implemented to the individuals from the control group who are willing to have the program.

Randomization Step 1: Randomization Method The names of the pregnant women admitted to the high-risk pregnancy service are written by the service nurse to the patient's hospitalization list according to the hospitalization dates. In order to differentiate the experimental and control groups, a notebook with the order of hospitalization from 1 to 80 was prepared by the researcher considering that there may be losses. The differentiation of the experimental and control groups was carried out by a simple random sampling method. The numbers that will be entered into the sample were determined by generate number www.random.org. Then, the women who met the criteria for inclusion in the sample were recorded in the notebook according to the order of hospitalization by the nurse in charge of in the high-risk pregnancy service. The numbers determined according to randomized numbers in the hospitalization book were adjusted to be the order of hospitalization. The experimental, and control groups were determined according to the order of hospitalization.

The numbers that make up the experimental, and control group are as follows; Experimental group: 1, 2, 3,4, 7, 8, 9, 11, 14, 21, 22, 24, 25, 26, 27, 29, 31, 37, 39, 41, 42, 45, 46, 48, 51, 52, 53, 54, 56, 57, 59, 60, 62, 65, 67, 68, 70,71, 74, 79 Control group: 5, 6, 10, 12, 13, 15, 16, 17, 18, 19, 20, 23, 28, 30, 32, 33, 34, 35, 36, 38, 40, 43, 44, 47, 49, 50, 55, 58, 61, 63, 64, 66, 69, 72, 73, 75, 76, 77, 78, 80 Step 2: Concealing the randomization data The separation of the experimental and control group was carried out by a third person as the nurse in charge of the service who had no association with the research. The service nurse in charge wrote the names of the hospitalized women in a notebook prepared by the researcher in accordance with the order of hospitalization. The notebook included no data about the numbers which belong to the experimental or control groups. The woman involved in the study was directed to the researcher by the nurse in charge with the envelope involving the number of the women.

Step 3: Practice The researcher found out the number of the patient after opening the envelope. From the numbers previously determined for the experimental and control group, the researcher included the women to the experimental or control group.

Step 4: Masking (Blinding) The women included in the sample of the study do not know which group they are involved in. The data of the experimental and control group was also hidden from the staff of the clinic. One by one interviews were performed in order to prevent the women from contacting each other in the experimental, and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Pregnants >24 weeks <34 weeks hospitalized in the high-risk pregnancy service of the relevant hospital,
* Speaking Turkish,
* Being literate,
* Be over 18 years old
* Being primigravida,
* At least 2 days have passed since admission to the service

Exclusion Criteria:

* Pregnants <24 weeks >34 weeks hospitalized in the high-risk pregnancy service of the relevant hospital,
* Not being willing to participate in the study,
* Having a diagnosed psychiatric illness.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Information Form | To both group at baseline ( before intervention)
  In the form prepared by the researcher in line with the literature review, ıt is a structured form consisting of closed-ended questions in order to determine individual characteristics such as, the age of the pregnant women, the number of pregnancies, the number of living children, social support resources, concomitant medical and psychiatric diseases, etc.
Depression, Anxiety and Stress Scale (DASS-21) | To both group at baseline ( before intervention)
  DAS-21 was created by Lovibond and Lovibond as an abbreviation of DAS-42. The validity and reliability study of the Turkish version of the "Depression Anxiety Stress-21 (DAS-21) scale in normal and clinical samples" was conducted by Sarıçam (2018). In the normal sample, it was found to be 0.85 for the depression subscale, 0.80 for the anxiety and 0.77 for the stress, respectively. For the clinical sample, it was 0.87 for depression, 0.85 for anxiety and 0.81 for stress. This scale is a 4-point Likert-type scale and consists of seven questions each measuring "depression, stress and anxiety dimensions". Getting 5 points or more from the depression sub-dimension, 4 points or more from anxiety, and 8 points or more from stress indicates that the individual has a related problem.
Depression, Anxiety and Stress Scale (DASS-21) | To both group immediately after the intervention
  DAS-21 was created by Lovibond and Lovibond as an abbreviation of DAS-42. The validity and reliability study of the Turkish version of the "Depression Anxiety Stress-21 (DAS-21) scale in normal and clinical samples" was conducted by Sarıçam (2018). In the normal sample, it was found to be 0.85 for the depression subscale, 0.80 for the anxiety and 0.77 for the stress, respectively. For the clinical sample, it was 0.87 for depression, 0.85 for anxiety and 0.81 for stress. This scale is a 4-point Likert-type scale and consists of seven questions each measuring "depression, stress and anxiety dimensions". Getting 5 points or more from the depression sub-dimension, 4 points or more from anxiety, and 8 points or more from stress indicates that the individual has a related problem.
Depression, Anxiety and Stress Scale (DASS-21) | To both group postpartum 4-6 week
  DAS-21 was created by Lovibond and Lovibond as an abbreviation of DAS-42. The validity and reliability study of the Turkish version of the "Depression Anxiety Stress-21 (DAS-21) scale in normal and clinical samples" was conducted by Sarıçam (2018). In the normal sample, it was found to be 0.85 for the depression subscale, 0.80 for the anxiety and 0.77 for the stress, respectively. For the clinical sample, it was 0.87 for depression, 0.85 for anxiety and 0.81 for stress. This scale is a 4-point Likert-type scale and consists of seven questions each measuring "depression, stress and anxiety dimensions". Getting 5 points or more from the depression sub-dimension, 4 points or more from anxiety, and 8 points or more from stress indicates that the individual has a related problem.
Depression, Anxiety and Stress Scale (DASS-21) | To both group postpartum 3 month
  DAS-21 was created by Lovibond and Lovibond as an abbreviation of DAS-42. The validity and reliability study of the Turkish version of the "Depression Anxiety Stress-21 (DAS-21) scale in normal and clinical samples" was conducted by Sarıçam (2018). In the normal sample, it was found to be 0.85 for the depression subscale, 0.80 for the anxiety and 0.77 for the stress, respectively. For the clinical sample, it was 0.87 for depression, 0.85 for anxiety and 0.81 for stress. This scale is a 4-point Likert-type scale and consists of seven questions each measuring "depression, stress and anxiety dimensions". Getting 5 points or more from the depression sub-dimension, 4 points or more from anxiety, and 8 points or more from stress indicates that the individual has a related problem.
Psychological Well-Being Scale : | To both group at baseline ( before intervention)
  It was developed by Diener et al. (2009) to measure socio-psychological well-being as a complement to existing measures of well-being. The items of the scale, which was adapted into Turkish by Telef (2013) and whose validity and reliability studies were conducted, are answered between 1 and 7, as I strongly disagree (1) to I strongly agree (7). The scale has a single factor structure and the Cronbach alpha coefficient is 0.80. All items are expressed positively. Scores range from 8 (strongly disagree to all items) to 56 (strongly agree to all items). A high score indicates that the person has many psychological resources and strengths. Although the scale does not provide individual measures of well-being, it does provide an overview of positive functioning in different areas believed to be important.
Psychological Well-Being Scale : | To both group immediately after the intervention
  It was developed by Diener et al. (2009) to measure socio-psychological well-being as a complement to existing measures of well-being. The items of the scale, which was adapted into Turkish by Telef (2013) and whose validity and reliability studies were conducted, are answered between 1 and 7, as I strongly disagree (1) to I strongly agree (7). The scale has a single factor structure and the Cronbach alpha coefficient is 0.80. All items are expressed positively. Scores range from 8 (strongly disagree to all items) to 56 (strongly agree to all items). A high score indicates that the person has many psychological resources and strengths. Although the scale does not provide individual measures of well-being, it does provide an overview of positive functioning in different areas believed to be important.
Psychological Well-Being Scale : | To both group postpartum 4-6 week
  It was developed by Diener et al. (2009) to measure socio-psychological well-being as a complement to existing measures of well-being. The items of the scale, which was adapted into Turkish by Telef (2013) and whose validity and reliability studies were conducted, are answered between 1 and 7, as I strongly disagree (1) to I strongly agree (7). The scale has a single factor structure and the Cronbach alpha coefficient is 0.80. All items are expressed positively. Scores range from 8 (strongly disagree to all items) to 56 (strongly agree to all items). A high score indicates that the person has many psychological resources and strengths. Although the scale does not provide individual measures of well-being, it does provide an overview of positive functioning in different areas believed to be important.
Psychological Well-Being Scale : | To both group postpartum 3 month
  It was developed by Diener et al. (2009) to measure socio-psychological well-being as a complement to existing measures of well-being. The items of the scale, which was adapted into Turkish by Telef (2013) and whose validity and reliability studies were conducted, are answered between 1 and 7, as I strongly disagree (1) to I strongly agree (7). The scale has a single factor structure and the Cronbach alpha coefficient is 0.80. All items are expressed positively. Scores range from 8 (strongly disagree to all items) to 56 (strongly agree to all items). A high score indicates that the person has many psychological resources and strengths. Although the scale does not provide individual measures of well-being, it does provide an overview of positive functioning in different areas believed to be important.
Intolerance of uncertainty scale | To both group at baseline ( before intervention)
  The Intolerance of Uncertainty Scale was developed by Carleton et al. (2007). The scale was adapted to Turkish culture by Sarıçam et al. (2014). The scale has 12 items designed in the form of a five-point Likert scale. The scale has two sub-dimensions (future-oriented anxiety and debilitating anxiety) and a total score can be taken from the scale. The general internal consistency coefficient of the Intolerance of Uncertainty Scale is 0.88. Sample items of the scale; "Unexpected events bother me so much", "I have to stay away from all uncertain situations" (Sarıçam et al., 2014).
Intolerance of uncertainty scale | To both group immediately after the intervention
  The Intolerance of Uncertainty Scale was developed by Carleton et al. (2007). The scale was adapted to Turkish culture by Sarıçam et al. (2014). The scale has 12 items designed in the form of a five-point Likert scale. The scale has two sub-dimensions (future-oriented anxiety and debilitating anxiety) and a total score can be taken from the scale. The general internal consistency coefficient of the Intolerance of Uncertainty Scale is 0.88. Sample items of the scale; "Unexpected events bother me so much", "I have to stay away from all uncertain situations" (Sarıçam et al., 2014).
Intolerance of uncertainty scale | To both group postpartum 4-6 week
  The Intolerance of Uncertainty Scale was developed by Carleton et al. (2007). The scale was adapted to Turkish culture by Sarıçam et al. (2014). The scale has 12 items designed in the form of a five-point Likert scale. The scale has two sub-dimensions (future-oriented anxiety and debilitating anxiety) and a total score can be taken from the scale. The general internal consistency coefficient of the Intolerance of Uncertainty Scale is 0.88. Sample items of the scale; "Unexpected events bother me so much", "I have to stay away from all uncertain situations" (Sarıçam et al., 2014).
Intolerance of uncertainty scale | To both group postpartum 3 month
  The Intolerance of Uncertainty Scale was developed by Carleton et al. (2007). The scale was adapted to Turkish culture by Sarıçam et al. (2014). The scale has 12 items designed in the form of a five-point Likert scale. The scale has two sub-dimensions (future-oriented anxiety and debilitating anxiety) and a total score can be taken from the scale. The general internal consistency coefficient of the Intolerance of Uncertainty Scale is 0.88. Sample items of the scale; "Unexpected events bother me so much", "I have to stay away from all uncertain situations" (Sarıçam et al., 2014).
Edinburgh Postnatal Depression Scale (EPDS) | To both group postpartum 4-6 week
  The Edinburgh Postpartum Depression Scale was developed by Cox in 1987. The scale aims to screen postpartum depression in women. The most widely used screening instrument for perinatal depression in both international and Turkish research.The validity and reliability study of the scale in our country was conducted by Engindeniz (1996). The scale consists of 10 items. Items are evaluated in a 4-point Likert format and scored between 0-3. The lowest score that can be obtained from the scale is 0, and the highest score is 30. The cut-off point of the scale is calculated as 12. Individuals who score above this score are considered as a risk group for depression.
Edinburgh Postnatal Depression Scale (EPDS) | To both group postpartum 3 month
  The Edinburgh Postpartum Depression Scale was developed by Cox in 1987. The scale aims to screen postpartum depression in women. The most widely used screening instrument for perinatal depression in both international and Turkish research.The validity and reliability study of the scale in our country was conducted by Engindeniz (1996). The scale consists of 10 items. Items are evaluated in a 4-point Likert format and scored between 0-3. The lowest score that can be obtained from the scale is 0, and the highest score is 30. The cut-off point of the scale is calculated as 12. Individuals who score above this score are considered as a risk group for depression.
Program Evaluation and Satisfaction Survey | Experimental group immediately after the intervention
  The questionnaire to be applied to pregnant women who participated in the cognitive-behavioral approach-based stress reduction program applied to high-risk pregnants aims to measure the satisfaction level of the participants. This form, prepared by the researcher for the intervention group, contains closed-ended questions and will be applied after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sevil Yılmaz, Assit.Prof., Study Director — Istanbul University-Cerrahpasa Florence Nightingale Nursing Faculty
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)